CLINICAL TRIAL: NCT01184612
Title: Motivational Interviewing Delivered by Existing Prison Staff: A Randomized Controlled Study of Effectiveness on Substance Use After Release
Brief Title: Effects of Motivational Interviewing in Prison
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: the research committee of the National Prison and Probation Administration (Unknown)
Responsible Party: Lars Forsberg Ph D, Karolinska institutet
Allocation: Randomized | Masking: Single | Purpose: Treatment
Other Study IDs: 30225613
Record Dates: First submitted 2010-08-18; First posted 2010-08-19 (Estimated); Last update posted 2010-08-19 (Estimated); Status verified 2003-10

CONDITIONS: Alcohol Abuse
Keywords: Inmates with heavy use of alcohol or drugs
MeSH Terms: conditions — Alcoholism | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- (BSF) MI sessions (Active Comparator): 5 semi-structured manualised MI sessions was conducted by existing prison staff having undergone 3 days of Motivational Interviewing workshop training and 2 days of training with the BSF manual.
  Interventions: Behavioral: Motivational Interviewing; MI
- (BSF+) MI sessions with supervision (Active Comparator): 5 semi-structured manualised MI sessions was conducted by ordinary prison staff having undergone 3 days of Motivational Interviewing workshop training and 2 days of training with the BSF manual, followed by ongoing Motivational Interviewing training with feedback based on audio taped sessions in peer supervision groups.
  Interventions: Behavioral: Motivational Interviewing; MI
- (UPI) Usual Planning Interview (Active Comparator): 5 sessions was conducted by prison staff according to usual working practices, with the exception that content was structured into 5 sessions and audio recorded. The provision of a government decree served as a basis for the intervention, covering planning of prison activities and post release arrangements including strategies for drug use cessation.
  Interventions: Behavioral: Motivational Interviewing; MI

INTERVENTIONS:
Behavioral: Motivational Interviewing; MI — MI is a communication style defined as a collaborative, person-centred form of guiding to elicit and strengthen motivation to change. The method is based on four principles: showing empathy; developing discrepancy between the subject's current behaviour and an alternate, more desired, behaviour; reinforcing self-efficacy; and "rolling" with resistance to change. Client arguments for change are elicited and reinforced in an atmosphere that is empathic, collaborative and supportive of autonomy. The choice to change and the responsibility for change remain with the client.

SUMMARY:
Motivational Interviewing (MI) is a communication style demonstrated to decrease drug and alcohol use. A five session MI intervention (BSF) was implemented in the Swedish correctional system. The intervention was delivered by counsellors with workshop only MI training (BSF) or by counsellors with workshop MI training followed by peer group supervision based on audio taped feedback (BSF+).

Aim was to examine whether BSF in prisons reduces drug and alcohol use more effectively than interviews conducted according to the usual planning interview routine (UPI).

ELIGIBILITY:
Inclusion Criteria:

* Born between 01-01-1954 and 31-12-1984;
* Conditional release no later than 30-06-2005 (this was extended to 19-09-2005 and again to 31-03-2006);
* Swedish or Norwegian speaker;
* Not having previously received BSF in remand or any other prison;
* Heavy use of alcohol or drugs, measured by the standard prison and probation system: 1= occasional use; 2= heavy use;
* ASI interview at intake;
* No order for deportation after release from prison

Exclusion Criteria:

-

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 296 (Actual)
Dates: Start 2004-04; Primary Completion 2007-03 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
number of days with substance use | of the last 30 days
  alcohol- or drug use as measured by the Addiction Severity Index (ASI) at intake and at 10 months after release

SECONDARY OUTCOMES:
reported days of illegal activity | during the preceding 30 days
  as measured by Addiction Severity Index at intake and 10 months after release
number of days working | during the last 30 days
  as measured by the Addiction Severity Index at intake and 10 months after release

CONTACTS AND LOCATIONS:
Overall Officials: Lars G Forsberg, Ph D, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Dep Clin Neuroscience, Stockholm, Sweden